CLINICAL TRIAL: NCT01387321
Title: A Study of BYL719 in Adult Patients With Advanced Solid Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CBYL719X1101
Record Dates: First submitted 2011-06-27; First posted 2011-07-04 (Estimated); Last update posted 2020-12-08 (Actual); Status verified 2018-08

CONDITIONS: Advanced Solid Tumor
Keywords: Pi3K; Advanced solid tumor
MeSH Terms: interventions — Alpelisib

ARMS (1):
- BYL719 (Experimental)
  Interventions: Drug: BYL719

INTERVENTIONS:
Drug: BYL719

SUMMARY:
In this study, BYL719 will be administered to adult patients with advanced solid tumors whose disease has progressed despite standard therapy or for whom no standard therapy exists. The trial will investigate the safety and tolerability and determine the MTD of BYL719 in Japanese patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically-confirmed, advanced unresectable solid tumors Availability of a representative formalin fixed paraffin embedded tumor tissue sample
* At least one measurable or non-measurable lesion Age ≥ 18 years
* Eastern Cooperative Oncology Group(ECOG) Performance Status ≤ 2 Good organ (hepatic, kidney, BM) function at screening/baseline visit

Exclusion Criteria:

* Brain metastasis unless treated and free of signs/symptoms attributable to brain metastasis in the absence of corticosteroid therapy and anti-epileptic therapy.
* Prior treatment with PI3K inhibitor
* Patient with peripheral neuropathy NCI-CTC Grade ≥ 2
* Patient with diarrhea NCI-CTC Grade ≥ 2
* Patient with acute or chronic pancreatitis
* Impaired cardiac function or clinically significant cardiac disease incl unstable angina pectoris ≤ 3 months prior to starting study drug and Acute Myocardial Infarction (AMI) ≤ 3 months prior to starting study drug
* Patients with clinically manifest diabetes mellitus, history of gestational diabetes mellitus or documented steroid-induced diabetes mellitus
* Women who are pregnant or breast feeding or adults of reproductive potential not employing an effective method of birth control

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2011-09-22 (Actual); Primary Completion 2015-11-25 (Actual); Study Completion 2015-11-25 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose | 4 Weeks

SECONDARY OUTCOMES:
Safety assessed by type, frequency and severity of adverse events | 4 Months
  Patients may continue treatment with BYL719 until the patient experiences unacceptable toxicity or progressive disease, an expected average of 4 months.
Efficacy assessed by RECIST | 4 months
  Patients may continue treatment with BYL719 until the patient experiences unacceptable toxicity or progressive disease, an expected average of 4 months.
  RECIST - Response Evaluation Criteria In Solid Tumors
To characterize the PK Profiles (AUC, Cmax, Tmax, CL/F, Vz/F, T1/2) | 4 months
  Patients may continue treatment with BYL719 until the patient experiences unacceptable toxicity or progressive disease, an expected average of 4 months.
Levels of biomarkers in tumor and skin | 4 months
  Patients may continue treatment with BYL719 until the patient experiences unacceptable toxicity or progressive disease, an expected average of 4 months.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (3):
- Japan (3):
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Chuo-ku, Tokyo
  - Novartis Investigative Site, Koto-ku, Tokyo

REFERENCES:
- See also: Results for CBYL719X1101 can be found on the Novartis Clinical Trials Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=15347